CLINICAL TRIAL: NCT04693039
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerance and Pharmacokinetics of Phenlarmide Tablets in Patients With Parkinson's Disease in the Early and Middle Stages
Brief Title: Study on the Safety, Tolerance and Pharmacokinetics of Phenlarmide Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shijiazhuang Yiling Pharmaceutical Co. Ltd (Industry)
Collaborators: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: FLZPD1003
Record Dates: First submitted 2020-12-28; First posted 2021-01-05 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- FLZ-150mg (Experimental): Drug：Phenlarmide；Dosage：150mg；
  Interventions: Drug: Phenlarmide
- FLZ-300mg (Experimental): Drug：Phenlarmide；Dosage：300mg；
  Interventions: Drug: Phenlarmide
- FLZ-600mg (Experimental): Drug：Phenlarmide；Dosage：600mg；
  Interventions: Drug: Phenlarmide
- FLZ-900mg (Experimental): Drug：Phenlarmide；Dosage：900mg；
  Interventions: Drug: Phenlarmide
- Placebo-150mg (Placebo Comparator): Drug：Placebo；Dosage：150mg；
  Interventions: Drug: Placebo
- Placebo-300mg (Placebo Comparator): Drug：Placebo；Dosage：300mg；
  Interventions: Drug: Placebo
- Placebo-600mg (Placebo Comparator): Drug：Placebo；Dosage：600mg；
  Interventions: Drug: Placebo
- Placebo-900mg (Placebo Comparator): Drug：Placebo；Dosage：900mg；
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Phenlarmide — Dosage form：Tablet; Give the medicine once a day，4 weeks is a cycle of administration, a total of 3 cycles of administration.
  Other Names: FLZ-150mg; FLZ-300mg; FLZ-600mg; FLZ-900mg
  Arms: FLZ-150mg; FLZ-300mg; FLZ-600mg; FLZ-900mg
Drug: Placebo — Dosage form：Tablet; Give the medicine once a day，4 weeks is a cycle of administration, a total of 3 cycles of administration.
  Other Names: Placebo-150mg; Placebo-300mg; Placebo-600mg; Placebo-900mg
  Arms: Placebo-150mg; Placebo-300mg; Placebo-600mg; Placebo-900mg

SUMMARY:
1. To evaluate the safety and tolerability of Phenlarmide tablets in patients with Parkinson's disease in the early and middle stages.
2. To evaluate the pharmacokinetics of Phenlarmide tablets in patients with Parkinson's disease.
3. To explore the efficacy of Phenlarmide tablets in the treatment of early and mid-term Parkinson's disease.

DETAILED DESCRIPTION:
1. Objective to evaluate the tolerance and safety of multiple administration of fenloramide tablets in patients with early and mid-term Parkinson's disease: To evaluate the adverse events of DLT and MTD, adverse reactions, clinical laboratory tests (blood routine, blood biochemistry, coagulation function, urine routine, stool routine), vital signs, 12 lead ECG and physical examination of fenloramide tablets in patients with early and mid-term Parkinson's disease .
2. Objective to evaluate the pharmacokinetics of fenloramide tablets in patients with Parkinson's disease in early and middle stages. The main PK parameters included Tmax, SS, Cmax, SS, cavg, SS, Ke, T1 / 2, Cl / F (only fenloramide prototype), VZ / F (only fenloramide prototype), auc0-24, SS, aucinf, SS, auc0 last, SS, AUC_ %Extrap, DF, etc.
3. Objective to explore the efficacy of fenloramide tablets in the treatment of early and mid-term Parkinson's disease, and to observe the changes of UPDRS and CGI.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and sign the informed consent, understand the research process and requirements, and volunteer to participate in the study;
2. over 30 years old and have no gender limit;
3. Patients diagnosed with Parkinson's disease according to the Chinese diagnostic criteria for Parkinson's disease (2016 Edition);
4. Hoehn-Yahr grade ≤ 3;
5. The Unified Parkinson's disease scale (UPDRS) motor score (Part III) ≥ 10;
6. Not using anti Parkinson's disease drugs within 28 days before enrollment;
7. If the subjects are receiving dopamine receptor agonists (such as Pramipexole, etc.), anticholinergic drugs (such as Benzhexol Hydrochloride, etc.), monoamine oxidase B (MAO-B) inhibitors (such as Selegiline, Rasagiline, etc.), and N-methyl-D-aspartate (NMDA) receptor antagonists (such as Amantadine), they should stop using the drugs 28 days before the screening period;
8. Patients who had been treated with levodopa preparation (including levodopa compound preparation) for less than 6 months before screening, and had not received levodopa preparation treatment within 28 days before screening period.

Exclusion Criteria:

1. Atypical Parkinson's symptoms due to the use of drugs (such as Flunarizine, Metoclopramide), nervous system diseases, genetic metabolic diseases, encephalitis, cerebrovascular diseases or other degenerative diseases (such as progressive supranuclear paralysis);
2. Patients with dementia, active mental illness or hallucination, severe depression (Beck Depression Scale - Ⅱ ≥ 29 points at screening), or Mini-Mental State Examination (MMSE) < 25 points;
3. Those who have received neurosurgical operation or electrical stimulation (such as pallidotomy, thalamotomy, deep brain electrical stimulation, etc.);
4. Patients with clinically significant abnormal liver function were defined as total bilirubin > 1.5 times of the upper limit of normal value or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 times of the upper limit of normal value;
5. Patients with clinically significant renal dysfunction: creatinine clearance rate (CCR) < 30 ml / min (using Cockcroft-Gault formula);
6. Patients with uncontrollable or severe cardiovascular diseases, including NYHA grade II or above congestive heart failure, unstable angina pectoris, myocardial infarction, arrhythmia requiring treatment at the time of screening, and QTc interval prolongation more than 480ms, in 6 months before the first administration of trial drug;
7. There is a history of heart, liver, kidney, respiratory, digestive, endocrine, immune or blood system diseases considered by researchers to be serious;
8. During the screening period, the patients with HIV positive, HBV or HCV infection and syphilis infection were active;
9. Patients with malignant tumor within 5 years before screening were excluded from cervical carcinoma in situ, skin basal cell or squamous cell carcinoma, local prostate cancer after radical operation and breast intraductal carcinoma in situ after radical operation;
10. There were significant food or drug allergy history or hypersensitivity reaction judged by researchers as having clinical significance;
11. Participants in any clinical trials within 3 months before administration of the study;
12. Pregnant or lactating women, or those whose serum hCG test is positive before trial administration, who are unable or unwilling to take contraceptive measures approved by the researcher during the study period and within 3 months after the end of the study according to the instructions of the researcher;
13. Those considered unsuitable by the researchers to participate in this clinical trial.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
the dose limiting toxicity (DLT) | through study completion, an average of 6 months
  The occurrence of Dose limiting toxicity.
Tmax, ss | through study completion, an average of 6 months
  After administration, the time when the highest concentration of drug appeared in plasma
Efficacy evaluation | through study completion, an average of 6 months
  explore the efficacy of fenolamide tablets in the treatment of early and middle stage Parkinson's disease, and observe the changes of UPDRS and CGI.
maximum tolerable dose (MTD) | through study completion, an average of 6 months
  The occurrence of Maximum tolerable dose.
adverse events | through study completion, an average of 6 months
  The occurrence rate of adverse events.
adverse reactions | through study completion, an average of 6 months
  The occurrence rate of adverse reactions
blood routine | through study completion, an average of 6 months
  Check whether the red blood cell system, white blood cell system and platelet system are normal
blood biochemistry | through study completion, an average of 6 months
  The contents of various ions, sugars, lipids, proteins, enzymes, hormones and metabolites in blood were detected
coagulation function | through study completion, an average of 6 months
  Four coagulation parameters including prothrombin time (PT), activated partial thromboplastin time (APTT), thrombin time (TT) and fibrinogen (FIB) were evaluated.
urine routine | through study completion, an average of 6 months
  Urine routine examination includes urine color, transparency, pH, red blood cells, white blood cells, epithelial cells, tube type, protein, specific gravity and urine sugar.
stool routine | through study completion, an average of 6 months
  Routine stool tests include the detection of red and white blood cells in feces, bacterial sensitivity test, occult blood test (OB) and inspection of eggs.
Body temperature | through study completion, an average of 6 months
  One of the vital signs.
12 lead ECG | through study completion, an average of 6 months
  Evaluation of QT interval
Blood pressure | through study completion, an average of 6 months
  Assess whether systolic blood pressure and diastolic blood pressure are normal.
Heart rate | through study completion, an average of 6 months
  One of the vital signs.
Breathing | through study completion, an average of 6 months
  Assess if breathing is normal
Cmax, ss | through study completion, an average of 6 months
  The highest concentration of the drug in the plasma after administration
Cavg, ss | through study completion, an average of 6 months
  The quotient of the area under the plasma concentration time curve divided by the interval time within a dose interval after the plasma concentration reaches the steady state.
Ke | through study completion, an average of 6 months
  The ratio of the amount of compound eliminated from the body to the total amount in the body in unit time
t1/2 | through study completion, an average of 6 months
  The time required for the concentration of a drug to drop by half in an organism
CL/F (fenoxamide prototype only) | through study completion, an average of 6 months
  The amount of a substance excreted by the kidney per minute
Vz/F (fenoxamide prototype only) | through study completion, an average of 6 months
  After the drug reaches dynamic equilibrium in the body, the ratio of the drug dose in the body to the blood concentration is called the apparent distribution volume
AUC0-24, ss | through study completion, an average of 6 months
  After administration, the area under the 0-24 hour time curve of blood concentration absorbed into human circulation
AUCinf, ss | through study completion, an average of 6 months
  After administration, the area under the time curve of 0-infinity of the blood concentration absorbed into human circulation
AUC0-last，ss | through study completion, an average of 6 months
  After administration, the area under the time curve of 0-the last accurately determined sample collection time of the blood concentration absorbed into human circulation
AUC_%Extrap | through study completion, an average of 6 months
  the area under the curve that has been derived after extrapolation of Residual Area
DF | through study completion, an average of 6 months
  The index reflecting the unbalanced situation of transportation in time

CONTACTS AND LOCATIONS:
Overall Officials: biao chen, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Chen Biao, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No